CLINICAL TRIAL: NCT06783218
Title: An Integrative Study of the Role of the Microbiome, Metabolome, Transcriptome and Chronobiology in the Context of Type 2 Diabetes.
Brief Title: An Integrative Study of the Role of Microbiome, Metabolome, Transcriptome and Chronobiology in the Context of Type 2 Diabetes.
Acronym: KRONODIABET
Status: Completed | Type: Observational
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Collaborators: European Union Next Generation (Unknown); Ministry of Science and Innovation, Spain (Other Government); Government of Navarra (Unknown); CIBER de Fisiopatología de la Obesidad y Nutrición (CIBERobn). (Unknown)
Responsible Party: Sponsor
Other Study IDs: KRONODIABET
Record Dates: First submitted 2024-12-18; First posted 2025-01-20 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2024-12

CONDITIONS: Prediabetes / Type 2 Diabetes; Obesity and Overweight; Insulin Resistance
Keywords: prediabetes; type 2 diabetes; obesity; microbiome; metabolome; eating behaviour; circadian rhythm; glycaemic control
MeSH Terms: conditions — Prediabetic State; Diabetes Mellitus, Type 2; Obesity; Overweight; Insulin Resistance; Feeding Behavior

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Whole blood, serum, plasma, white cells, saliva, faeces
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Prediabetes/type 2 diabetes: Individuals with excess weight (overweight or obesity) and drug-naïve prediabetes or type 2 diabetes.
- Controls: Invididuals without glycaemic control impairment and normal weight, matched on sex and age with the prediabetes/type 2 diabetes group.

SUMMARY:
The goal of this descriptive clinical study is to investigate daily oscillations in glycaemic control between healthy adults and adults with excess weight and who have early-stage prediabetes or T2D and are not taking medications for glycaemic control. The study also explores how these differences relate to changes in daily patterns in oral microbiome and metabolome, circadian markers, and lifestyle factors such as eating, physical activity, light exposure and appetite.

The main questions to answer are:

1. Do adults with excess weight and prediabetes/T2D exhibit a disruption of the circadian system compared to healthy individuals? If so, are these disruptions manifested in hormone levels, gene expression, microbiota composition and function, metabolite levels and appetite regulation?
2. Does chrono-disruption contribute to the dysregulation of glucose metabolism and responses to lifestyle factors in individuals with excess weight and prediabetes/T2D?

Researchers will compare two groups:

* Healthy adults with normal weight.
* Adults with excess weight (overweight or obesity) with prediabetes/T2D who are not on diabetes medications.

The study will involve both semi-controlled settings (where food intake and physical activity are controlled) and free-living conditions.

Participants will:

* Wear devices: Use a continuous glucose monitor and a circadian monitoring device for 14 days.
* Attend clinical visits: Visit the Nutritional Intervention Unit (NIU) 4 times for body composition measurements, sample collection (blood, saliva a faeces) and to answer questionnaires. .
* Participate in a 12.5-hours clinical visit day in the NIU under semi-controlled conditions, with the purpose of collecting blood samples before and after breakfast and saliva samples every 4 hours, covering a full 24-hour cycle.
* Keep track of daily habits: Maintain their usual lifestyle while keeping a food diary and recording appetite related feelings.

DETAILED DESCRIPTION:
Compelling evidence suggests that type 2 diabetes (T2D) can often be prevented by adopting healthy lifestyle. However, current standard recommendations may not fully account for individual differences, limiting their effectiveness. Factors such as genetics and daily lifestyle patterns influence how individuals respond to these recommendations. For example, disrupted sleep patterns or irregular eating schedules can make it difficult to maintain healthy habits, ultimately affecting blood glucose control. Such disruptions are associated with disturbances in the body's internal clock, also known as circadian rhythms. In this sense, chrono-disruption (i.e., disruption of circadian rhythms) has been shown to impair glucose metabolism. Individuals at high risk of T2D are characterized by loss of diurnal rhythmicity in the insulin oscillatory pattern. Similarly, recent studies suggest that disruptions in daily fluctuations of hormone levels, gene expression, microbiota composition, and metabolite profiles are associated with poorer blood glucose control.

The present project relies on the hypothesis that individuals with excess weight and drug-naïve prediabetes or type 2 diabetes, compared to healthy individuals, exhibit a disruption of the circadian system. This is manifested by loss in daily oscillations and altered oscillatory patterns across multiple physiological processes, including hormone production, gene expression, microbiota composition and function, and metabolite composition and secretion. Chrono disruption contributes to the dysregulation of glucose metabolism, changes in appetite regulation and response to external cues and, consequently, impaired glycaemic control in this population.

The Kronodiabet study is a 2-week observational study with two parallel study groups, matched by age and gender, according to the following conditions: adults with overweight or obesity and impaired glucose metabolism (drug-naive prediabetes or type 2 diabetes); and adults with normal weight and no alterations in glucose metabolism.

Experimental design: Each participant, once recruited, will attend the NIU at the Center for Nutrition Research of the University of Navarra on 4 occasions. At visit 1 (V1), participants will come to the NIU and will be fitted with a continuous glucose monitoring sensor and a circadian monitoring device, which will be worn during the main study visit (V2) and the following 12 ± 2 full days (field period phase) and body composition will be analysed through dual energy x-ray absorptiometry (DEXA). At this visit (V1), participants will bring a stool sample collected no later than 48 hours prior to arrival at the NIU. In visit 2 (V2), lasting 12 hours and 30 minutes, participants will arrive to the NIU (where the entire visit will take place) after at least 8 hours of fasting. During this visit, participants will be provided with the meals to be consumed throughout the day and blood draws and completion of questionnaires will be carried out. In addition, 4 out of the 7 saliva samples required for the analysis of the oral microbiota, metabolome and gene and hormone determination will be collected every 4 hours. The remaining saliva samples (3/7) will be collected at home, until the 24-hour period is completed. On the following day (V3), participants will come back to the NIU to deliver the samples collected at home. In addition, they will be given the necessary material for the field study period. During the field phase (which will last 2 weeks) participants will be asked not to change their habitual lifestyle, including diet, exercise and timing. In the final visit (V4), body composition measurements will be taken and the circadian and glucose monitoring sensors and completed questionnaires will be collected, concluding the study.

The specific objectives are:

1. To characterize the phenotype, behavioral traits and lifestyle habit, as well as the microbiome, metabolome and transcriptome in healthy individuals and individuals with overweight/obesity and drug-naïve prediabetes/type 2 diabetes.
2. To investigate, under free-living conditions, daily oscillations in glycaemia, food behavior and circadian parameters of the main circadian synchronizers.
3. To compare daily oscillations in oral microbiota and metabolome, along with daily oscillations of circadian markers, under semi-controlled conditions, between healthy individuals and individuals with overweight/obesity and drug-naïve prediabetes/type 2 diabetes.
4. To study, from an integrated perspective, daily oscillations in glycemic control, through the integration of omics (metagenomics, metabolomics), clinical and lifestyle data, in the absence and presence of excess weight and impaired glucose metabolism.

ELIGIBILITY:
Inclusion Criteria (T2D group):

* Women and men between the ages of 30 and 70.
* Meet any criteria diagnosis of prediabetes or type 2 diabetes according to the American Diabetes Association (ADA), without pharmacological treatment for glycaemic control.
* Excess weight, according to body mass index (BMI) value > 25 kg/m2.
* Body fat percentage, measured by bioelectrical impedance analysis (BIA), above the normal range, according to age and sex, following the classification from Gallagher D, et al. Am J Clin Nutr. 2000;72(3):694-701.

Inclusion Criteria (Healthy group):

* Women and men between the ages of 30 and 70.
* No impaired glucose metabolism according to ADA diagnostic criteria
* Normal weight, according to BMI value (18,5 - 24,9 kg/m2)
* Body fat percentage, measured by BIA, within the normal range, according to age and sex, following the classification from Gallagher D, et al. Am J Clin Nutr. 2000;72(3):694-701.

Exclusion Criteria:

* Chronotype within the categories "extreme evening" (<34) or "extreme morning" (>76), according to the Hörne-Orberg Morning-Evening Questionnaire (MEQ) classification.
* Weight changes (± 4.5 kg) during the last 3 months.
* Habitually consuming ≥ 14 units of alcohol/week in women and ≥ 21 units of alcohol/week in men.
* Self-reported use of drugs of abuse in the last 12 months.
* Be an active smoker or have quit smoking within the last 3 months.
* Night or late shift work (finishing later than 11 pm on a permanent basis).
* Recent travel across 2 or more time zones during the last month before the start of the study.
* Show poor cooperation or, in the opinion of the investigator, have difficulty following the study procedures.
* In the case of women, being pregnant or breastfeeding .
* Blood donation in the 3 months prior to the beginning of the study.

Medical conditions:

* Oral diseases, inflammation or lesions at the time of the study.
* Any clinical condition, including chronic metabolic diseases, systemic intestinal, hepatic or renal diseases, when the research team consider that it may influence the results of the study.
* Severe hyperlipidaemia, severe hypertension or hypothyroidism, untreated or treated for less than 3 months with stable dose.
* Have relevant functional or structural abnormalities of the digestive tract, such as malformations, angiodysplasias, active peptic ulcers, chronic inflammatory diseases or malabsorption.
* Subjects who have undergone surgery of the digestive tract with permanent sequelae, including surgical treatment for obesity.
* Any type of psychological/psychiatric impairment such as depressive pathology, anxiety or bipolar disorder, when the research team consider that it may influence the results of the study.
* Any type of cancer or be undergoing treatment for it, or that a period of at least 5 years has not elapsed since its eradication.
* A diagnosed eating disorder (such as bulimia or binge eating disorder)
* Presence of any type of health problem that may affect sleep
* Any infection at the time of the study, especially respiratory or intestinal infection.

Medication:

* Be under continuous pharmacological/hormonal treatment that may affect glycaemic control.
* Current or within the previous 2 months use of prescription or non-prescription medication or nutritional supplements that have the potential to affect glycaemic control, as well as biochemical analyses. For food supplements containing biotin, they are permitted provided that their consumption is omitted 48 h before blood draws.
* Current or within the previous 2 months use of nutritional supplements or prescription or non-prescription drugs that may affect the microbiota (probiotics, prebiotics, fibre, antibiotics, antifungals).
* Taking any medication that may seriously affect circadian rhythms (melatonin receptor agonist drugs (tasimelteon, ramelteon), drugs for the treatment of drowsiness (modafinil, armodafinil), or with sedative effects (benzodiazepines, zolpidem)) or nutritional supplements that contain melatonin and are likely to affect circadian rhythms, except if on a stable dose for 3 months or more.
* Cholesterol-lowering medication, except if on a stable dose for 3 months or more.
* Blood pressure lowering medication, unless on a stable dose for 3 months or more.
* Medication that may affect appetite and body weight (e.g. antidepressants, thyroid) unless on a stable dose for 3 months or more and without significant side effects.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals from a region in the north of Spain. People registered in the Nutrition Research Centre's own database will be invited. In addition, other recruitment channels will be used, such as flyers, advertisements in local press, medical centres and hospitals, social networks and websites.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2024-03-21 (Actual); Primary Completion 2024-10-15 (Actual); Study Completion 2024-10-28 (Actual)

PRIMARY OUTCOMES:
Percentage coefficient of variation of intra-day glucose levels (%CV) | Clinical Investigation Day 2 (24-hours)
  Measured by continuous glucose monitoring sensor during semi-controlled conditions in the main clinical investigation day (%)

SECONDARY OUTCOMES:
Glycaemic variation | 14 days
  Measured by continuous glucose monitor (FreeStyle Libre Pro, Abbott)
Glycated haemoglobin (HbA1c) | Screening, Clinical Investigation Day 2
  Blood samples, reported in % and in mmol/mol. For screening purposes, HbA1c will also be determined using capillary blood samples at the screening visit.
Fasting serum glucose | Screening, Clinical Investigation Day 2
  Serum samples, reported in mg/dl
Postprandial serum glucose | Clinical Investigation Day 2, blood samples taken every 30 min for 2 hours (4 timepoints in total)
  Serum samples, reported in mg/dl, collected every 30 minutes for 2 hours after consuming breakfast. iAUC will be calculated including blood sample collected at baseline.
Fasting serum insulin | Clinical Investigation Day 2
  Serum samples, reported in mU/L, determined by ELISA
Postprandial serum insulin | Clinical Investigation Day 2, blood samples taken every 30 min for 2 hours (4 timepoints in total)
  Serum samples, reported in mU/L, collected every 30 minutes for 2 hours after consuming breakfast, determined by ELISA. iAUC will be calculated including blood sample collected at baseline.
Fasting serum Peptide C | Clinical Investigation Day 2
  Serum samples, reported in ng/mL, determined by ELISA
Homeostasis Model Assessment for Insulin Resistance (HOMA-IR) | Clinical Investigation Day 2
  Calculated as (fasting basal insulin (mU/mL) x fasting glucose (mg/dL)/405
Fasting serum total cholesterol | Clinical Investigation Day 2
  Serum samples, reported in mg/dL
Fasting serum HDL cholesterol | Clinical Investigation Day 2
  Serum samples, reported in mg/dL
Fasting serum LDL cholesterol | Clinical Investigation Day 2
  Calculated using Friedewald's equation: total cholesterol - (triglycerides/5) - HDL-cholesterol
Fasting serum triglycerides | Clinical Investigation Day 2
  Serum samples, reported in mg/dL
Postprandial serum triglycerides | Clinical Investigation Day 2, blood samples taken every 30 min for 2 hours (4 timepoints in total)
  Serum samples, reported in mg/dL, collected every 30 minutes for 2 hours after consuming breakfast. iAUC will be calculated including blood sample collected at baseline.
Fasting serum alanine aminotransferase (ALT) | Clinical Investigation Day 2
  Fasting serum samples, reported in U/L
Fasting serum aspartate aminotransferase (AST) | Clinical Investigation Day 2
  Fasting serum samples, reported in U/L
Fasting serum gamma-glutamyl transferase (GGT) | Clinical Investigation Day 2
  Fasting serum samples, reported in U/L
Triglyceride-glucose index (TyG index) | Clinical Investigation Day 2
  Calculated using the following equation: Ln [(fasting triglycerides) (mg/dL) x fasting glucose (mg/dL)] / 2
Fatty Liver Index (FLI) | Clinical Investigation Day 2
  Calculated using the following equation: (e0.953×loge(triglycerides)+0.139×BMI+0.718×loge(GGT)+0.053×waistcircumference-15.745)/ (1 + e0.953×loge(triglycerides)+0.139×BMI+0.718×loge(GGT)+0.053×waistcircumference-15.745) × 100.
Fasting serum/plasma glucagon-like peptide-1 (GLP-1) | Clinical Investigation Day 2
  Serum/plasma samples, reported in pmol/L, determined by ELISA
Postprandial serum/plasma glucagon-like peptide-1 (GLP-1) | Clinical Investigation Day 2, blood samples taken every 30 min for 2 hours (4 timepoints in total)
  Serum/plasma samples, reported in pmol/L, collected every 30 minutes for 2 hours after consuming breakfast, determined by ELISA. iAUC will be calculated including blood sample collected at baseline.
Fasting serum/plasma ghrelin | Clinical Investigation Day 2
  Serum/plasma samples, reported in pmol/L
Postprandial serum/plasma ghrelin | Clinical Investigation Day 2, blood samples taken every 30 min for 2 hours (4 timepoints in total)
  Serum/plasma samples, reported in pmol/L, collected every 30 minutes for 2 hours after consuming breakfast, determined by ELISA. iAUC will be calculated including blood sample collected at baseline.
Fasting serum/plasma leptin | Clinical Investigation Day 2
  Serum/plasma samples, reported in ng/mL
Hemogram | Clinical Investigation Day 2
  Blood samples collected at fasting state
Daily rhythms of wrist temperature fragmentation | Clinical Investigation Day 2 (24-hours) and 14 days (field phase)
  Wrist temperature will be measured using a circadian monitoring device (Kronowise 3.0) and the circadian parameter fragmentation will be calculated as intradaily variability.
Daily rhythms of wrist temperature regularity | Clinical Investigation Day 2 (24-hours) and 14 days (field phase)
  Wrist temperature will be measured using a circadian monitoring device (Kronowise 3.0) and the circadian parameter regularity will be calculated as interdaily stability.
Daily rhythms of wrist temperature amplitude | Clinical Investigation Day 2 (24-hours) and 14 days (field phase)
  Wrist temperature will be measured using a circadian monitoring device (Kronowise 3.0) and the circadian parameter amplitude will be calculated as relative amplitude and normalised relative amplitude.
Daily rhythms of circadian light exposure | Clinical Investigation Day 2 (24-hours) and 14 days (field phase)
  Circadian light exposure intensity, expressed as lux, will be measured using a circadian monitoring device (Kronowise 3.0)
Daily rhythms of visible light exposure | Clinical Investigation Day 2 (24-hours) and 14 days (field phase)
  Visible light exposure intensity, expressed as lux, will be measured using a circadian monitoring device (Kronowise 3.0)
Daily rhythms of activity | Clinical Investigation Day 2 (24-hours) and 14 days (field phase)
  Activity, measured as acceleration, will be determined using a circadian monitoring device (Kronowise 3.0)
Daily rhythms of time in movement | Clinical Investigation Day 2 (24-hours) and 14 days (field phase)
  Time in movement will be determined using a circadian monitoring device (Kronowise 3.0)
Integrated variable TAP (Temperature, Motor activity, Body Position) | Clinical Investigation Day 2 (24-hours) and 14 days (field phase)
  TAP will be determined by integrating three simultaenous recordings: skin wrist temperature (T), motor activity (A) and body position (P) from a circadian monitoring device (Kronowise 3.0) to determine individual circadian system status (i.e., chronotype)
Baseline and change from baseline in body weight at the end of the study | Clinical Investigation Day 2 (week 0) and Clinical Investigation Day 4 (week 2)
  Measured by bioimpedance and reported in kg
Height | Screening (V0) and Clinical Investigation Day 1 (V1)
  Measured by stadiometer and reported in m
Baseline and change from baseline in body mass index at the end of the study | Clinical Investigation Day 2 (week 0) and Clinical Investigation Day 4 (week 2)
  Body mass index will be calculated as follows: weight (kilograms)/(height (m)*height (m)), and expressed as kg/m2
Baseline and change from baseline in body fat at the end of the study | Clinical Investigation Day 2 (week 0) and Clinical Investigation Day 4 (week 2)
  Measured by bioimpedance and DXA (only at baseline) and reported in kg and percentage.
Baseline and change from baseline in body fat-free mass at the end of the study | Clinical Investigation Day 2 (week 0) and Clinical Investigation Day 4 (week 2)
  Measured by bioimpedance and DXA (only at baseline) and reported in kg.
Baseline and change from baseline in lean mass at the end of the study | Clinical Investigation Day 2 (week 0) and Clinical Investigation Day 4 (week 2)
  Measured by bioimpedance and DXA (only at baseline) and reported in kg.
Baseline and change from baseline in body water at the end of the study | Clinical Investigation Day 2 (week 0) and Clinical Investigation Day 4 (week 2)
  Measured by bioimpedance and reported in kg.
Baseline and change from baseline in waist circumference at the end of the study | Clinical Investigation Day 2 (week 0) and Clinical Investigation Day 4 (week 2)
  Measured in fasting condition using a measuring tape and reported in centimeters
Baseline and change from baseline in hip circumference at the end of the study | Clinical Investigation Day 2 (week 0) and Clinical Investigation Day 4 (week 2)
  Measured in fasting condition using a measuring tape and reported in centimeters
Baseline and change from baseline in visceral fat level at the end of the study | Clinical Investigation Day 2 (week 0) and Clinical Investigation Day 4 (week 2)
  Measured in fasting condition by bioimpedance and expressed as level (from 0 to 40).
Android adipose tissue | Clinical Investigation Day 1 (V1)
  Determined by DXA and expressed as percentage of total body fat and fat mass in grams.
Gynoid adipose tissue | Clinical Investigation Day 1 (V1)
  Determined by DXA and expressed as percentage of total body fat and fat mass in grams.
Gynoid lean tissue | Clinical Investigation Day 1 (V1)
  Determined by DXA and expressed as percentage of total lean mass and lean mass in grams.
Android lean tissue | Clinical Investigation Day 1 (V1)
  Determined by DXA and expressed as percentage of total lean mass and lean mass in grams.
Ratio trunk/total fat mass | Clinical Investigation Day 1 (V1)
  Determined by DXA and calculated as the ratio of trunk fat to total body fat.
Ratio legs/total fat mass | Clinical Investigation Day 1 (V1)
  Determined by DXA and calculated as the ratio of legs fat to total body fat.
Visceral adipose tissue volume and mass | Clinical Investigation Day 1 (V1)
  Determined by DXA and expressed as volume, in cm3, and mass, in grams.
Salivary cortisol determinations | Clinical Investigation Day 2 (V2); saliva samples taken every four hour for 24 hours (7 time points in total)
  Saliva samples shall be collected every 4 hours for 24 hours, starting at 8 a.m. in the laboratory and ending at 8 a.m. the following day at home. Samples shall be collected by active salivation using a sample collection device, which contains a cotton swab.
Salivary melatonin determinations | Clinical Investigation Day 2 (V2); saliva samples taken every four hour for 24 hours (7 time points in total)
  Saliva samples shall be collected every 4 hours for 24 hours, starting at 8 a.m. in the laboratory and ending at 8 a.m. the following day at home. Samples shall be collected by active salivation using a sample collection device, which contains a cotton swab.
Oscillations in the expression of clock genes in saliva | Clinical Investigation Day 2 (V2); saliva samples taken every four hour for 24 hours (7 time points in total)
  Saliva samples shall be collected every 4 hours for 24 hours, starting at 8 a.m. in the laboratory and ending at 8 a.m. the following day at home. Samples shall be collected by passive drainage using a sample collection device, which contains a RNA/DNA preservative. Gene expression analyses will be performed by Real Time Polymerase Chain Reaction (RT-PCR) and quantified as relative expression compared to housekeeping genes.
Oral microbial community composition rhythmicity | Clinical Investigation Day 2 (V2); saliva samples taken every four hour for 24 hours (7 time points in total)
  Saliva samples shall be collected every 4 hours for 24 hours, starting at 8 a.m. in the laboratory and ending at 8 a.m. the following day at home. Samples shall be collected by passive drainage using a sample collection device, which contains a RNA/DNA preservative. Shotgun sequencing/16S sequencing will be performed for the metagenomic analysis and microbiota rhythmicity will be investigated.
Oral metabolite rhythmicity | Clinical Investigation Day 2 (V2); saliva samples taken every four hour for 24 hours (7 time points in total)
  Saliva samples shall be collected every 4 hours for 24 hours, starting at 8 a.m. in the laboratory and ending at 8 a.m. the following day at home. Samples will be collected by active salivation using a sample collection device, which contains a cotton swab. Oral metabolome profile will be assessed by broad-spectrum, untargeted metabolomics.

OTHER OUTCOMES:
Chronotype as assessed by Morningness-Eveningness Questionnaire (MEQ) | At screening
  The MEQ score classifies individuals according to their chronotype. Scores can range from 16 to 86 points. Scores of 41 or less indicate 'evening type'.
  Scores of 59 or more indicate 'morning type'. Scores between 42-58 indicate 'intermediate type'.
Chronotype as assessed by Munich Chronotype Questionnaire (MCTQ) | Clinical Investigation Day 2 (V2)
  The MCTQ uses the midpoint between sleep on- and offset on free days (mid-sleep on free days, MSF) to assess chronotype.
Subjective appetite sensations | Clinical Investigation Day 2 (V2) (during 14 hours; immediately before and 1.5 and 3 h after every meal, 15 time points in total) and during 3 non-consecutive days during the field phase (free-living conditions; immediately before and after every meal)
  Scores using a 100 mm Visual Analogue Scales (VAS) will be used to assess subjective appetite sensatios. A combined appetite score will be calculated and AUC at 4h for the Clinical Investigation Day 2 (V2) and on the three days of dietary recording during the field phase, following the trapezoid method, will be calculated.
Food cravings as assesed by the Control of Eating Questionnaire | Clinical Investigation Day 2 (V2) (at baseline) and 7 days after V2, during the field-phase
  Craving control, sweet cravings, salty cravings and positive mood scores will be assessed using a 100 mm visual analogue scales. Participants will be asked to respond based on overall feelings over the past 7 days.
Baseline eating pattern as assessed by Frequency of Consumption Questionnaire (FFQ) | Clinical Investigation Day 2 (V2)
  A validated 137-item semi-quantitative FFQ to assess individual's habitual food intake
Self-reported sleep quality as assessed by the Pittsburgh Sleep Quality Index (PSQI) | Clinical Investigation Day 2 (V2)
  Self-administered questionnaire that assess qualitative and quantitative aspects of sleep quality (subjective quality, latency, duration, habitual efficiency, disturbances, hypnotic use and daytime dysfunction)
Self-reported quality of life as assessed by the SF-12 | Clinical Investigation Day 2 (V2)
  Self-administered questionnaire that qualitatively measures self-perceived health status and health-related quality of life.
Faecal microbiota profile | Up to 48 hours before Clinical Investigation Day 2 (V2) (1 time point)
  Stool samples shall be collected no later than 48 hours before day 2 of the clinical investigation. After DNA extraction, metagenomic analysis will be performed by 16S rRNA gene sequencing.
Serum metabolite profile | Clinical Investigation Day 2 (V2)
  Identification and quantification of metabolites in serum samples collected in a fasting state will be performed. Serum metabolome profile will be assessed by broad-spectrum, untargeted metabolomics.
Transcriptome profiling in peripheral blood | Clinical Investigation Day 2 (V2)
  Blood samples will be collected at fasting state. RNA-seq will be performed for gene expression and characterisation of functional pathways in peripheral blood.
Socio-demographic and individual characteristics from an interview with the research staff | At screening
  Socio-demographic aspects will be asked for descriptive purposes, including age, sex, nationality, education level, civil status and work status. Additionally, medical history and use of medication and nutritional supplements will be asked.
Self-reported energy intake | 3 non-consecutive days during the field phase (free-living conditions), of which one will be a weekend day.
  The average total dietary intake over 3 days will be calculated as: ((day1 + day2)/2 x 5 + day3x2)/7), where day 1 and 2 are the food intake for working days and day 3 are the food intake for a weekend day
Self-reported macronutrient intake | 3 non-consecutive days during the field phase (free-living conditions), of which one will be a weekend day.
  The average total dietary intake over 3 days will be calculated as: ((day1 + day2)/2 x 5 + day3x2)/7), where day 1 and 2 are the food intake for working days and day 3 are the food intake for a weekend day
Self-reported daily eating window | 3 non-consecutive days during the field phase (free-living conditions), of which one will be a weekend day.
  Eating occasions will be defined as the consumption of >25 kcal, and will be used to calculate the daily eating window
Self-reported energy density | 3 non-consecutive days during the field phase (free-living conditions), of which one will be a weekend day.
  Average total amount and percentage of total daily calories consumed in each of the intakes of the day as well as the energy density of the diet for each of the 3 days, excluding caloric beverages (water, diet drinks) will be calculated. Energy density will be calculated as follows: day1 (kJ or kcal)/ day1 (g).
Presence of risky eating behaviours as assessed by the Eating Attitudes Test 26 (EAT-26) | Clinical Investigation Day 2 (V2)
  Total score is the sum of the scores of the 26 items of the scale. The items are answered on a 4-point Likert-type scale (0=never to 3=always). A score above 20 indicates a potential risk for behavioral eating disorder.
Presence of risky eating behaviors as assessed by Three Factor Eating Questionnaire (TFEQ) | Clinical Investigation Day 2 (V2)
  TFEQ assess eating behavior thourgh a score defines three dimensions of human eating behaviour, including food restraint, disinhibition and hunger)
Presence of risky eating behaviours as assessed by the Problem Eating Behavior Questionnaire (PEBQ) | Clinical Investigation Day 2 (V2)
  It consists of a score and 1 open-ended question that assesses the presence of eating behaviours potentially implicated in obesity. A qualitative examination will be carry out.

CONTACTS AND LOCATIONS:
Overall Officials: Pedro González-Muniesa, PhD, Principal Investigator — Center for Nutrition Research. University of Navarra; María Jesús Moreno-Aliaga, PhD, Principal Investigator — Center for Nutrition Research. University of Navarra; Ana Velasco-Andonegui, MSc, Study Chair — Center for Nutrition Research. University of Navarra
Locations (1):
- Center for Nutrition Research. University of Navarra, Pamplona, Navarre, Spain

IPD SHARING:
Plan to Share IPD: No